CLINICAL TRIAL: NCT02762643
Title: An Open-label, Randomized, Crossover Study to Evaluate the Pharmacokinetics and Safety of a Fixed Dose Combination of Raloxifen/Cholecalciferol Compared With Coadministration of Raloxifen and Cholecalciferol in Healthy Male Subjects
Brief Title: DP-R213 Pharmacokinetics Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alvogen Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DP-CTR213-I-01
Record Dates: First submitted 2016-04-29; First posted 2016-05-05 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Healthy
Keywords: DP-R213
MeSH Terms: interventions — Raloxifene Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RT group (Experimental): combination dose of Raloxifene and Cholecaliferol and DP-R213 in order
  Interventions: Drug: DP-R213; Drug: Raloxifene; Drug: Cholecaliferol
- TR group (Experimental): combination dose of Raloxifene and Cholecaliferol and DP-R213 in order
  Interventions: Drug: DP-R213; Drug: Raloxifene; Drug: Cholecaliferol

INTERVENTIONS:
Drug: DP-R213 — Investigational product is prescribed to all of randomized subjects
Drug: Raloxifene — Investigational product is prescribed to all of randomized subjects
Drug: Cholecaliferol — Investigational product is prescribed to all of randomized subjects

SUMMARY:
A randomized, open-label, crossover, Phase I clinical trial to compare the pharmacokinetics of DP-R213 (Raloxifenel and Cholecaliferol fixed dose combinations) in comparison to each component administered alone in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* IBW ±20%
* signed the informed consent form prior to the study participation

Exclusion Criteria:

* Clinically significant disease
* Previously donate whole blood within 2 months or component blood within 1 month
* Clinically significant allergic disease
* Taken IP in other trial within 3 months
* An impossible one who participates in clinical trial by investigator's decision including laboratory test result

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-05; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | up to 96 hours post dose
Peak Plasma Concentration (Cmax) | up to 96 hours post dose

IPD SHARING:
Plan to Share IPD: No